CLINICAL TRIAL: NCT05455515
Title: The GISE-ShockCalcium Registry - An Investigator Driven Italian All Comers Registry of Calcified Lesions Treated With Intravascular Lithotripsy
Brief Title: The GISE (Società Italiana di Cardiologia Interventistica) - ShockCalcium Registry
Status: Recruiting | Type: Observational
Sponsor: Fondazione GISE Onlus (Other)
Collaborators: Shockwave Medical, Inc. (Industry); INNOVA HTS SRL (Unknown); University of Padova (Other)
Responsible Party: Sponsor
Other Study IDs: GISE_Shockcalcium
Record Dates: First submitted 2022-05-20; First posted 2022-07-13 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-03

CONDITIONS: Coronary Disease
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: IVL procedures — Intravascular Lithotripsy (IVL)

SUMMARY:
The GISE-SHOCKCALCIUM Registry is an Investigator Driven Italian All Comers prospective, observational, multicenter Italian IVL registry of Calcified lesions Treated with Intravascular Lithotripsy. The main purpose is to evaluate the efficacy and safety of coronary lithotripsy for treatment of severe calcified lesion. A total of 2000 patients with coronary calcified lesions will be enrolled in 24 months. The registry will be conducted in approximately 50 interventional cardiology centers in Italy with at least 2 IVL procedures per 24 months. Primary endpoint: Target lesion failure (TLF) at 1 year.

Secondary safety endpoints: in Hospital Target lesion failure (TLF); Target Lesion Failure at 30 days; definite or probable stent thrombosis; procedural angiographic safety endpoints. Secondary effectiveness endpoints: device crossing and IVL delivery success; angiographic success; QCA (quantitative coronary angiography) outcome; Imaging outcome.

DETAILED DESCRIPTION:
This is a prospective, observational, multicenter Italian IVL registry designed to evaluate the efficacy and safety of coronary lithotripsy for treatment of severe calcified lesion.

This registry is planned to be conducted at approximately 30-50 sites in Italy and to include a total of 2000 patients with coronary calcified lesions.

The Principal Investigators will approach all the Italian centers with at least 2 IVL procedures per month via the regional GISE Coordinator and based on the IVL volume of the various hospitals with IVL in the previous 18 months (excluding the period February-June 2020). Possible regulatory or budgetary constrictions expected to limit future application of IVL will also be considered. Centers should be approached by on-line questionnaires and during regional teleconferences to agree to collect data for all IVL procedures, fill a screening log for all calcified lesions, perform a complete clinical 1 year follow-up of all IVL patients, including collection of source documents for event adjudication. Participation in OCT (optical coherence tomography) or IVUS (Intravascular UltraSound) sub-studies (clinically mandated imaging) will be highly encouraged agreeing to perform documented pull-backs across the calcified treated/stented segment and provide images for off-line analysis from a central core laboratory.

The registry will consist of 3 essential parts: a screening period (patient and lesion selection), a treatment period (PCI with IVL lesion preparation and stent implantation), and a follow-up period (1 year).

Patients will be screened, according to the flowchart and stratified at baseline by angiographic evaluation or intravascular imaging.

Patients will be scheduled to undergo an intracoronary lithotripsy procedure using an appropriately sized Shockwave catheter (Shockwave Medical, Fremont, CA).

All arteries with visible calcium with the appearance of facing lines in at least one view will be included in the registry. In calcified lesions with questionable indications (not too long/thick angiographically) the use of IVUS or OCT will be strongly encouraged, but final selection will be left at the Investigators' preference. IVUS should be used instead of OCT in the presence of CKD (chronic kidney disease) and for very distal or aorto-ostial stenoses, all relative or absolute contraindications for OCT.

Selection of additional devices (Rotablator, IVL, high pressure or cutting/scoring balloons) will also be performed at the Investigators' preference.

Lesions with angiographically severe calcification will be examined with QCA analysis and/or intravascular imaging in order to discriminate between lesions requiring direct treatment with IVL and lesions treatable with balloon pre-dilatation. IVL could be also performed in case of focal balloon under-expansion, defined as the persistence of a focal balloon indentation 28at a pressure of 16-18 Atm, in lesions with angiographically mild to moderate calcifications or no angiographically visible calcifications initially planned for conventional balloon pre-dilatation. Uncrossable lesions will receive RA (Rotablator atherectomy) as default strategy, with an option for IVL in case of suboptimal balloon expansion.

The sample size was estimated by considering the primary endpoint of the study, i.e., the comparison of the late (one year) composite endpoint of CV (cardiovascular) death, lesion-related MI (Myocardial infarction), TLF including clinically driven TLR (Target lesion revascularization), definite and probable ST (stent thrombosis) in IVL treatment compared to other interventions. A Monte Carlo (MC) simulation method was considered for the calculation. According to a sample size up to 2000 patients, a study size of 1900 patients for a 12% event ensures an average confidence interval length of 0.029 (Figure 4). The final sample size is 2000 adjusted for a 5% dropout rate.

ELIGIBILITY:
Inclusion Criteria:

* Patients is ≥ 18 years of age.
* Patients with calcified coronary artery disease requiring percutaneous revascularization with stent implantation who require an IVL with the Shockwave catheter.
* Presence of single or multiple calcifications at the lesion site defined by,

  a) angiography, with fluoroscopic radio-opacities noted without cardiac motion prior to contrast injection involving both sides of the arterial wall in at least one location and total length of calcium of at least 15 mm and extending partially into the target lesion, OR by b) IVUS or OCT, with presence of ≥270 degrees of calcium on at least 1 cross section
* Ability to tolerate dual antiplatelet agent (i.e. aspirin, clopidogrel, prasugrel, or ticagrelor for 1 year and single antiplatelet therapy for life)
* Ability to give written informed consent.
* Patient is able and willing to comply with all follow-up assessments

Exclusion Criteria:

* Refusal to participate in this study.
* Calcific lesion within a > 4 mm reference segment of the vessel
* Lesions in LIMA(left internal mammary artery)/RIMA (rightinternal mammary artery) or at the distal anastomosis of an SVG (saphenous vein grafts)
* All the usual relative contraindications to coronary angioplasty according to the clinical practice:
* Patient has active systemic infection
* Patient has a known untreated coagulation disorder
* Patient has allergy to imaging contrast media for which he/she cannot be pre-medicated
* Patient is pregnant or nursing
* Patients whose life expectancy is < 1 year
* Patients due to move abroad within 1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with coronary calcified lesions
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2022-09-17 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Primary composite safety endpoint: Target lesion failure (TLF): cardiovascular death | at 1 year
  Cardiovascular death defined as death resulting from cardiovascular causes:
  1. death caused by acute MI
  2. death caused by sudden cardiac arrest, including unwitnessed death
  3. death resulting from heart failure
  4. death caused by stroke
  5. death caused by cardiovascular procedures
  6. death resulting from cardiovascular hemorrhage
  7. death resulting from other cardiovascular cause
Primary composite safety endpoint: Target lesion failure (TLF): Target-vessel Myocardial infarction (TV-MI) | at 1 year
  based on CK-MB level >3x ULN with or without new pathologic Q-wave through discharge (peri-procedural MI) and using the 4th Universal Definition of MI beyond discharge
Primary composite safety endpoint: Target lesion failure (TLF): Target lesion revascularization (TLR) | at 1 year
  defined as a repeat percutaneous intervention of the target lesion or bypass surgery of the target vessel performed for restenosis or other complication of the target lesion, clinically or ischemia driven

SECONDARY OUTCOMES:
Secondary safety endpoints: in Hospital Target lesion failure (TLF) | at 1 year
  defined as a composite of cardiac death, target vessel related non-fatal myocardial infarction or need for unplanned target lesion revascularization
Secondary safety endpoints: Target lesion failure | at 30 days
  defined as a composite of cardiac death, target vessel related non-fatal myocardial infarction or need for unplanned target lesion revascularization
Secondary safety endpoints: Definite or probable stent thrombosis | at 1 year
  Definite stent thrombosis (ST) OR Pathological confirmation of ST determined by the evidence of recent thrombus within the stent at autopsy and/or examination of tissue retrieved following thrombectomy (visual/histology).
  Probable ST: Regardless of the time after the index procedure, any myocardial infarction that is related to documented acute ischemia in the territory of the implanted stent without angiographic confirmation of stent/scaffold thrombosis and in the absence of any other obvious cause)25.
  Timing of ST:
  Acute 0*-24h Subacute >24h-30day Late 30 day-1 year
  *0 is defined as the moment the patient is undraped and taken off the catheterization table25
Secondary safety endpoints: Procedural angiographic safety endpoints | at 1 year
  1. severe dissection: dissection in the target vessel greater than type B from National Heart, Lung, and Blood Institute classification
  2. coronary perforation defined as evidence of extravasation of dye or blood from the coronary artery during or following the interventional procedure. This is detected either by angiographic appearances consistent with dye outside of the vessel lumen or by echocardiographic evidence of a pericardial effusion.
  3. abrupt closure defined as an abrupt cessation of coronary flow to TIMI grade 0 or 1 flow before or at ≤5 mm distal to the lesion in an artery in which PTCA was attempted where there had previously been TIMI grade 2 or 3 flow prior to the procedure.
  4. slow flow or no-reflow: markedly delayed flow (TIMI grade 2 for slow flow, TIMI 0 or 1 for no reflow) in a target vessel with minimal (<30%) residual stenosis at the stented/scaffolded segment and no evidence of flow-limiting dissection
Secondary effectiveness endpoints: Device crossing and IVL delivery success | at 1 year
  defined by the ability to deliver the IVL catheter across the target lesion prior or after pre-dilatation and delivery of lithotripsy without serious arrhythmias during delivery or angiographic complications after IVL
Secondary effectiveness endpoints: Angiographic success | at 1 year
  Stent delivery with ≤30% residual stenosis and without serious angiographic complications

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Careggi Florence, Florence, Italy

IPD SHARING:
Plan to Share IPD: Undecided